CLINICAL TRIAL: NCT01594866
Title: A Double-blinded 6-week Prospective Study to Evaluate the Remission Rate According to Dose of Escitalopram (Lexapro®) in Patients With Major Depressive Disorder: a Preliminary Study
Brief Title: Lexapro®'s Efficacy After Dose Escalation in Remission Study
Acronym: LEADERS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Principal Investigator, Yong Min Ahn, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AYM-LEADERS
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder, remission, escitalopram
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram, 20mg, placebo (Placebo Comparator): escitalopram 20mg + placebo (same taste, appearance, texture of escitalopram 10mg)
  Interventions: Drug: escitalopram
- Escitalopram 20mg, escitalopram 10mg (Experimental): Escitalopram 20mg + Escitalopram 10mg
  Interventions: Drug: escitalopram

INTERVENTIONS:
Drug: escitalopram — escitalopram 20mg and 30mg p.o. daily, 6 weeks
  Other Names: Lexapro®
Drug: escitalopram — escitalopram 10mg p.o. for 1 week, and escitalopram 20mg p.o. for 3 weeks before randomized to placebo and experimental groups
  Other Names: Lexapro®

SUMMARY:
The purpose of this study is the evaluation of remission rate between escitalopram 20 mg and 30 mg in patients with major depressive disorder.

DETAILED DESCRIPTION:
In this study, the investigators are going to examine the efficacy of escitalopram after dose escalation and evaluate remission rate. This study design is the double-blinded 6-week prospective study. It would be useful for clinicians because there were few study of high-dose antidepressant treatment in lack of remission in major depressive disorder patients. To control of bias, the investigators included patients with lack of remission after 4-week escitalopram treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 ~ 65
* Patient with major depressive disorder according to DSM-IV criteria
* Patient have signed on the informed consent, and well understood the objective and procedure of this study.
* MADRS total score ≥ 18
* Competent patient who is manage to answer the questionnaires.
* In case of female at child-bearing age, consent to use appropriate contraceptive methods(oral pill, contraceptive injection, intrauterine device, double barrier method and contraceptive patch) during entire duration of this study.

Exclusion Criteria:

* In previous depressive episodes, no efficacy although more than one antidepressant treatment
* Allergy or hypersensitivity to escitalopram
* Diagnosed to schizophrenia or bipolar disorder or schizoaffective disorder (DSM-IV)
* MADRS 10 score ≥ 5, or patient who is supposed to be impossible to participate to this study due to clinical risk of suicide or aggressive behavior based on clinician's opinion
* Pregnant or breast-feeding female patient
* Significant biochemical or hematological abnormality or abnormal finding of urinalysis, based on clinician's opinion
* Significant severe medical condition
* Patients who take antipsychotics or mood stabilizer or other psychiatric drugs excluding benzodiazepines or beta blockers or hypnotics
* History of participating to other investigational drug trial within 1month prior to screening
* Investigator or employee at clinical trial center, personnel related to investigator or trial center on this or other study, or family of employee or investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | 6 weeks

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale-17 items (HAM-D) | 6 weeks
Hamilton Anxiety Rating Scale (HAM-A) | 6 weeks
Clinical Global Impression-severity (CGI-S) | 6 weeks
Clinical Global Impression-Improvement (CGI-I) | 6 weeks
Beck's Depression Inventory(BDI) | 6 weeks
WHO Quality Of Life scale Abbreviated Version(WHOQOL-BREF) | 6 weeks
Clinically Useful Depression Outcome Scale (CUDOS) | 6 weeks
Short From-36 Health survey (SF-36 Health survey) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yong Min Ahn, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea